CLINICAL TRIAL: NCT00094094
Title: Phase 2 Study of the Anti-Angiogenesis Agent AG-013736 as Second- or Later- Line Treatment in Patients With Advanced Non-Small Cell Lung Cancer
Brief Title: Anti-angiogenesis Agent AG-013736 in Patients With Advanced Non-Small Cell Lung Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Pfizer (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: A4061011
Record Dates: First submitted 2004-10-11; First posted 2004-10-14 (Estimated); Results first posted 2012-03-16 (Estimated); Last update posted 2012-06-26 (Estimated); Status verified 2012-06

CONDITIONS: Lung Neoplasms; Carcinoma, Non-small Cell Lung
MeSH Terms: conditions — Lung Neoplasms; Carcinoma, Non-Small-Cell Lung | interventions — Axitinib

ARMS (1):
- Axitinib (Experimental): AG-013736 is a vascular endothelial growth factor [VEGF] inhibitor
  Interventions: Drug: axitinib

INTERVENTIONS:
Drug: axitinib — Axitinib (AG-013736) tablet administered orally at a dose of 5 milligrams (mg) twice daily (BID) in cycles of 4 weeks.

SUMMARY:
This is a Phase 2 study being conducted at multiple centers in the United States and Germany. Patients having non-small cell lung cancer that has spread to other parts of the body (i.e., metastatic) or is locally advanced (i.e., Stage IIIB with malignant pleural effusion) are eligible to participate. Patients must have disease that has been treated with at least 1 prior treatment for metastatic disease (prior adjuvant treatment for localized disease does not count as prior treatment for metastatic disease). The purpose of the study is to test whether the angiogenesis inhibitor AG-013736 is an effective treatment for advanced non-small cell lung cancer as shown by the number of patients in the study who experience significant and durable tumor shrinkage

ELIGIBILITY:
Inclusion Criteria:

* Histologically documented non-small cell lung cancer with metastases (Stage IV or recurrent disease) or locally advanced (Stage IIIB) with malignant pleural effusion.
* At least 1 prior systemic therapy for metastatic disease (Prior adjuvant therapy for localized disease does not count as a prior therapy for metastatic disease).

Exclusion Criteria:

* Central lung lesions involving major blood vessels (arteries or veins). (Central lesions that maintain the structural integrity of vessels have the potential to bleed if the tumor lesion undergoes necrosis. MRI or CT angiography should be used in any case where there is any question as to whether blood vessels are involved.)
* Patients with a history of Grade 2 or worse hemoptysis are not eligible. Patients with a history of Grade 1 hemoptysis within 30 days of entry are not eligible

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2005-02; Primary Completion 2007-07 (Actual); Study Completion 2007-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (11):
- United States (10):
  - Pfizer Investigational Site, Irvine, California
  - Pfizer Investigational Site, Orange, California
  - Pfizer Investigational Site, Chicago, Illinois
  - Pfizer Investigational Site, Park Ridge, Illinois
  - Pfizer Investigational Site, Coon Rapids, Minnesota
  - Pfizer Investigational Site, Fridley, Minnesota
  - Pfizer Investigational Site, Robbinsdale, Minnesota
  - Pfizer Investigational Site, Charlotte, North Carolina
  - Pfizer Investigational Site, Nashville, Tennessee
  - Pfizer Investigational Site, Madison, Wisconsin
- Pfizer Investigational Site, Gauting, Germany

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A4061011&StudyName=Anti-angiogenesis%20Agent%20AG-013736%20in%20Patients%20with%20Advanced%20Non-Small%20Cell%20Lung%20Cancer

RESULTS

PARTICIPANT FLOW:
Groups:
- Axitinib: Axitinib (AG-013736) tablet administered orally at a dose of 5 milligram (mg) twice daily (BID) in cycles of 4 weeks. Treatment was administered continuously until progression or unacceptable toxicity occurred or the participant withdrew consent.
Period: Overall Study
Arm/Group | Axitinib
Started | 32
Completed | 0
Not Completed | 32
Not completed — Death | 2
Not completed — Lack of Efficacy | 23
Not completed — Adverse Event | 7

BASELINE CHARACTERISTICS:
Groups:
- Axitinib: Axitinib (AG-013736) tablet administered orally at a dose of 5 mg BID in cycles of 4 weeks. Treatment was administered continuously until progression or unacceptable toxicity occurred or the participant withdrew consent.
Arm/Group | Axitinib
Number analyzed (Participants) | 32
Age Continuous [Mean (Standard Deviation); unit: Years] | 64.1 (12.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13
  Male | 19

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Objective Response (OR)
Description: Percentage of participants with OR based assessment of confirmed complete response (CR) or confirmed partial response (PR) according to Response Evaluation Criteria in Solid Tumors (RECIST). Confirmed responses are those that persist on repeat imaging study at least 4 weeks after initial documentation of response. CR are defined as the disappearance of all lesions (target and/or non target). PR are those with at least 30 percent (%) decrease in the sum of the longest dimensions of the target lesions taking as a reference the baseline sum longest dimensions.
Time Frame: Baseline until the date of first documented progression or discontinuation from the study due to any cause, assessed every 8 weeks up to 98 weeks
Population: Study population included all participants who enrolled and received treatment.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Axitinib
Number analyzed (Participants) | 32
Percentage of participants | 9.4 [2.0 to 25.0]

2. Secondary Outcome: Progression-Free Survival (PFS)
Description: Time in days from start of study treatment to first documentation of objective tumor progression or death due to any cause. PFS was calculated as first event date minus the date of first dose of study medication plus 1. Tumor progression was determined from oncologic assessment data (where data meet the criteria for progressive disease [PD]), or from adverse event (AE) data (where the outcome was "Death").
Time Frame: Baseline until the date of first documented progression or death due to any cause, assessed every 8 weeks up to 98 weeks
Population: Study population included all participants who enrolled and received treatment.
Measure: Median (95% Confidence Interval); unit: Days
Arm/Group | Axitinib
Number analyzed (Participants) | 32
Days | 148 [109 to 213]

3. Secondary Outcome: Duration of Response (DR)
Description: Time in days from the first documentation of objective tumor response to objective tumor progression or death due to any cause. Duration of tumor response was calculated as the date of the first documentation of objective tumor progression or death due to cancer minus the date of the first CR or PR that was subsequently confirmed plus 1. DR was calculated for the subgroup of participants with a confirmed objective tumor response.
Time Frame: as for outcome 1
Population: Subgroup of participants from the study population with a confirmed objective tumor response (CR or PR).
Measure: Median (95% Confidence Interval); unit: Days
Arm/Group | Axitinib
Number analyzed (Participants) | 3
Days | 252 [179 to 322]

4. Secondary Outcome: Overall Survival (OS)
Description: Time in days from the start of study treatment to date of death due to any cause. OS was calculated as the death date minus the date of first dose of study medication plus 1. Death was determined from AE data (where outcome was death) or from follow-up contact data (where the participant current status was death). For participants who were alive, overall survival was censored at the last contact.
Time Frame: Baseline to death due to any cause or at least 1 year after the initial dose for the last treated participant
Population: Study population included all participants who enrolled and received treatment.
Measure: Median (95% Confidence Interval); unit: Days
Arm/Group | Axitinib
Number analyzed (Participants) | 32
Days | 450 [326 to NA] — Upper limit of confidence interval was not estimable due to the high number of participants censored for survival.

5. Other Pre Specified Outcome: Population Pharmacokinetics for Axitinib (AG-013736) Plasma Concentrations
Description: Population pharmacokinetic analysis involved mixed effects modeling using nonlinear mixed effects modeling (NONMEM) software. The intent of this analysis was to establish a basic population pharmacokinetic model for axitinib (AG-013736) and to determine inter-individual and residual variability in population (oral) clearance, and volume of distribution of drug. Relationship of demographic variables (gender, age, body weight, height and ethnicity), concomitant medications and measures of altered hepatic and renal function were examined by fitting measured axitinib (AG-013736) concentrations.
Time Frame: Day 1 (pre-dose), Day 29, Day 57 and then every 8 weeks up to 98 weeks
Population: Population pharmacokinetic values were not summarized as descriptive statistics since the data was not available for the single study and data for all the axitinib Phase 2 studies would be pooled together in a separate report.
Measure: Mean (Standard Deviation); unit: nanogram/milliliter (ng/mL)
Arm/Group | Axitinib
Number analyzed (Participants) | 0

6. Other Pre Specified Outcome: Plasma Concentrations of Soluble Proteins
Description: Plasma concentrations of soluble proteins (vascular endothelial growth factor [VEGF], placental growth factor [PlGF] and soluble vascular endothelial growth factor receptor-2 [sVEGFR2]) may be associated with tumor angiogenesis or tumor physiology and may correlate with efficacy or biological activity. It is presented as ratio to baseline, which is obtained by dividing the plasma soluble protein concentration at each time point by its concentration at baseline.
Time Frame: Day 1 (pre-dose) and then every 8 weeks up to 98 weeks
Population: Ratio to baseline values for plasma soluble proteins were not summarized as descriptive statistics since the data was not available for the single study and data for all the axitinib Phase 2 studies would be pooled together in a separate report.
Measure: Mean (Standard Deviation); unit: Ratio
Arm/Group | Axitinib
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Description: The same event may appear as both an AE and a SAE. However, what is presented are distinct events. An event may be categorized as serious in one subject and as nonserious in another subject, or one subject may have experienced both a serious and nonserious event during the study.
Arm/Group | Axitinib
Serious Adverse Events (participants affected / at risk) | 16/32
Other Adverse Events (participants affected / at risk) | 31/32
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Axitinib (N=32)
Acute coronary syndrome (Cardiac disorders) | 1
Bradycardia, not otherwise specified (NOS) (Cardiac disorders) | 1
Appendicitis (Gastrointestinal disorders) | 1
Colitis NOS (Gastrointestinal disorders) | 1
Diarrhoea haemorrhagic (Gastrointestinal disorders) | 1
Dysphagia (Gastrointestinal disorders) | 1
Large intestinal ulcer (Gastrointestinal disorders) | 1
Oesophageal stenosis acquired (Gastrointestinal disorders) | 1
Rectal haemorrhage (Gastrointestinal disorders) | 1
Disease progression NOS (General disorders) | 5
General physical health deterioration (General disorders) | 1
Bronchitis acute NOS (Infections and infestations) | 1
Infection NOS (Infections and infestations) | 1
Pneumonia NOS (Infections and infestations) | 1
Dehydration (Metabolism and nutrition disorders) | 2
Hyperkalaemia (Metabolism and nutrition disorders) | 1
Ataxia (Nervous system disorders) | 1
Cerebrovascular accident (Nervous system disorders) | 1
Convulsions NOS (Nervous system disorders) | 1
Transient ischaemic attack (Nervous system disorders) | 1
Confusion (Psychiatric disorders) | 3
Renal failure acute (Renal and urinary disorders) | 1
Chronic obstructive airways disease exacerbated (Respiratory, thoracic and mediastinal disorders) | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 1
Dyspnoea NOS (Respiratory, thoracic and mediastinal disorders) | 2
Dyspnoea exacerbated (Respiratory, thoracic and mediastinal disorders) | 1
Hypotension NOS (Vascular disorders) | 1
Inferior vena caval obstruction (Vascular disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Axitinib (N=32)
Anaemia (Blood and lymphatic system disorders) | 3
Tachycardia (Cardiac disorders) | 4
Hypothyroidism (Endocrine disorders) | 2
Abdominal pain (Gastrointestinal disorders) | 4
Abdominal pain upper (Gastrointestinal disorders) | 3
Constipation (Gastrointestinal disorders) | 6
Diarrhoea (Gastrointestinal disorders) | 15
Dyspepsia (Gastrointestinal disorders) | 7
Dysphagia (Gastrointestinal disorders) | 4
Flatulence (Gastrointestinal disorders) | 2
Glossodynia (Gastrointestinal disorders) | 3
Nausea (Gastrointestinal disorders) | 15
Oral discomfort (Gastrointestinal disorders) | 2
Oral pain (Gastrointestinal disorders) | 4
Stomatitis (Gastrointestinal disorders) | 2
Vomiting (Gastrointestinal disorders) | 10
Chest pain (General disorders) | 4
Fatigue (General disorders) | 27
Gait disturbance (General disorders) | 2
Mucosal inflammation (General disorders) | 5
Oedema peripheral (General disorders) | 5
Pain (General disorders) | 2
Bronchitis (Infections and infestations) | 2
Rhinitis (Infections and infestations) | 2
Upper respiratory tract infection (Infections and infestations) | 7
Traumatic haematoma (Injury, poisoning and procedural complications) | 2
Alanine aminotransferase increased (Investigations) | 2
Blood creatinine increased (Investigations) | 2
Weight decreased (Investigations) | 11
Degreased appetite (Metabolism and nutrition disorders) | 19
Dehydration (Metabolism and nutrition disorders) | 3
Hyperglycaemia (Metabolism and nutrition disorders) | 2
Hypoglycaemia (Metabolism and nutrition disorders) | 2
Hypokalaemia (Metabolism and nutrition disorders) | 4
Hypomagnesaemia (Metabolism and nutrition disorders) | 3
Hyponatraemia (Metabolism and nutrition disorders) | 4
Arthralgia (Musculoskeletal and connective tissue disorders) | 8
Back pain (Musculoskeletal and connective tissue disorders) | 3
Bone pain (Musculoskeletal and connective tissue disorders) | 2
Muscular weakness (Musculoskeletal and connective tissue disorders) | 5
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 4
Myalgia (Musculoskeletal and connective tissue disorders) | 3
Pain in extremity (Musculoskeletal and connective tissue disorders) | 4
Ataxia (Nervous system disorders) | 2
Dizziness (Nervous system disorders) | 3
Headache (Nervous system disorders) | 8
Neuropathy peripheral (Nervous system disorders) | 3
Somnolence (Nervous system disorders) | 2
Anxiety (Psychiatric disorders) | 2
Confusional state (Psychiatric disorders) | 2
Depression (Psychiatric disorders) | 2
Insomnia (Psychiatric disorders) | 4
Proteinuria (Renal and urinary disorders) | 6
Urinary retention (Renal and urinary disorders) | 2
Cough (Respiratory, thoracic and mediastinal disorders) | 11
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 12
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 10
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 4
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 3
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 2
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 2
Alopecia (Skin and subcutaneous tissue disorders) | 3
Dry skin (Skin and subcutaneous tissue disorders) | 3
Rash (Skin and subcutaneous tissue disorders) | 5
Rash erythematous (Skin and subcutaneous tissue disorders) | 2
Hypertension (Vascular disorders) | 10
Hypotension (Vascular disorders) | 2

LIMITATIONS AND CAVEATS:
Population pharmacokinetics and plasma concentrations of soluble proteins were not presented, as the data was not available for the single study and data for all the axitinib Phase 2 studies would be pooled together in a separate report.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.